CLINICAL TRIAL: NCT06678243
Title: Randomized Clinical Trial to Test the Efficacy of a Smartphone App for Smoking Cessation for Nondaily Smokers (SiS4)
Brief Title: Testing the mHealth App Intervention for Nondaily Smokers "SiS4"
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Bettina B. Hoeppner, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-501; 1R01CA282223 (NIH)
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-04

CONDITIONS: Smoking Cessation
Keywords: smoking; smartphone app; smoking cessation; QuitGuide; Smiling instead of Smoking; positive psychology; mHealth; nondaily smoking
MeSH Terms: conditions — Smoking Cessation; Smoking

STUDY DESIGN:
Intervention Model Description: single-blind, remote, randomized clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Smiling instead of Smoking (Experimental): Participants will be onboarded to the smartphone app "Smiling instead of Smoking" (SiS4) and will be asked to use it for 7 weeks while they quit smoking.
  Interventions: Behavioral: Smiling instead of Smoking
- QuitGuide (Active Comparator): Participants will be onboarded to the smartphone app "QuitGuide" (QG) which will be 're-branded', so that the name "Smiling instead of Smoking" will appear in the banner of the app instead of "QuitGuide", and will be asked to use it for 7 weeks while they quit smoking.
  Interventions: Behavioral: QuitGuide

INTERVENTIONS:
Behavioral: Smiling instead of Smoking — Participants randomized to the treatment condition will use the "Smiling instead of Smoking" (SiS) smartphone app. This app delivers and guides participants through two types of content to help them during their quit attempt: (1) positive psychology content (i.e., happiness habit-building exercises, happiness boost activity, and science-based information on the relevance of positive psychology activities) designed to help nondaily smokers maintain positive affect while they go through the process of smoking cessation; and (2) traditional behavioral smoking cessation content to guide their quit process based on US Clinical Practice Guidelines.
  Other Names: SiS4
  Arms: Smiling instead of Smoking
Behavioral: QuitGuide — Participants randomized to the control condition will use the National Cancer Institute (NCI)'s "QuitGuide" (QG) smartphone app. The QuitGuide app follows the US Clinical Practice Guidelines. The app is freely available on NCI's Smokefree.gov website, which is a recommended resource for treating smokers in the healthcare setting. The QuitGuide app is frequently used as a comparison app in smartphone app smoking cessation studies. It asks participants to set a quit day, track their mood and cravings, and log their cigarettes. It provides app users with guidance on quitting (i.e., "Learn to Quit" information), offers strategies to counter smoking triggers, and allows users to set reminders to stay smoke free (time and location based).
  Other Names: QG
  Arms: QuitGuide

SUMMARY:
The goal of this project is to test if a new behavioral treatment for people who smoke nondaily and wish to quit works. The new treatment is a smartphone app that engages users in positive psychology exercises and gives them tested tools for quitting smoking. The positive psychology exercises help users maintain their positive emotions while they quit smoking. This app has been developed with and for people who smoke nondaily through several steps of development.

The main questions it aims to answer are:

* Does the smoking cessation app (SiS4) help people who smoke nondaily quit smoking?
* How do people's attitudes towards smoking, their smoking urges, and their mental well-being shift when using the SiS4 app?

Researchers will compare the new app to an existing app that was developed for people who smoke daily to see if the new app works better to help people who smoke nondaily quit smoking.

Participants will:

1. Use a smartphone app every day for 7 weeks
2. Complete online surveys about their smoking, attitudes about smoking, withdrawal symptoms and smoking urges, app use, and mental well-being at enrollment as well as 2 weeks, 6 weeks, 3 months, 6 months and 12 months after the initially chosen quit date.

If the SiS4 app works well, it would be the first evidence-based quit-smoking treatment for people who smoke nondaily.

DETAILED DESCRIPTION:
The present study is a large-scale (n=1,600) single-blind, remote, parallel, randomized clinical trial (RCT) comparing our app, the SiS app, to the NCI's smartphone app "QuitGuide". The RCT will be conducted entirely remotely, because the app is intended to be accessible to smokers nationally without need for in person contact. All participants will set a targeted smoking cessation quit date and will be instructed to use the provided app for 7 weeks, 1 week prior to and 6 weeks post-quit. Online surveys will be conducted at enrollment and follow-up occurring 2 weeks, 6 weeks, 3 months, 6 months and 12 months after the initially chosen quit date. The primary outcome measure will be 30-day point-prevalence abstinence (PPA) at 6 months post-quit. The investigator team developed the app, "Smiling instead of Smoking (SiS)," specifically for and in collaboration with people who smoke less than daily. This app uses a positive psychology approach, in line with their preference to focus on positive self-identity and wellness.

The investigators have rigorously and iteratively developed and tested this app in a series of small scale prior studies. Study 1 (2017P001106) demonstrated feasibility and acceptability when smokers were onboarded in person. Study 2 (2018P002699) demonstrated feasibility and acceptability when smokers were onboarded remotely, nationwide. Study 3 (NCT04672239) demonstrated the app's ability to engage nondaily smokers and showed proof-of-concept efficacy in a small, randomized trial, where participants using the SiS app had significantly higher self-efficacy, lower craving, and higher positive affect at the end of treatment, compared to controls.

In this large-scale efficacy trial, the primary outcome measure will be 30-day point-prevalence abstinence (PPA) at 6-month post quit. The aims of the study are:

Aim 1: Test the effectiveness of the SiS app to improve smoking cessation outcomes

1. H1: 30-day PPA six months post quit will be higher for SiS compared to QuitGuide participants.
2. H2: SiS participants will have higher 30-day PPA at end of treatment and 12 months post quit.

Aim 2: Examine mechanisms and moderators of change

1. Using mediation modeling, the investigators will test if theorized mechanisms of change (i.e., self-efficacy, positive affect, or craving) account for observed effects on 30-day PPA six months post quit.
2. (Exploratory aim:) Using moderated mediation models, the investigators will examine if socioeconomic status, race, and/or the presence of mental health conditions moderate the effectiveness of SiS or moderate the mediation effects outlined in aim 2a.

Exploratory Aim 3: Explore app usage patterns and their relationship to smoking cessation

1. The investigators will identify patterns of overall app use, as identified by group-based trajectory modeling.
2. The investigators will conduct a feature-level analysis of the apps (i.e., which features got used how often).
3. The investigators will test if patterns of app use and/or feature use predict 30-day PPA six months post-quit.

If found to be efficacious, this study would provide the first evidence of an efficacious treatment (the SiS app) for people who smoke less than daily, for whom currently no treatment guidelines exist.

ELIGIBILITY:
* 18 years of age or older
* Sufficiently fluent in English to read and comprehend intervention and assessment materials
* Owns a smartphone (Android or iOS only)
* Currently smokes less than daily but at least weekly
* Has smoked 100+ cigarettes lifetime
* Has current intention to quit smoking
* Currently resides in the US
* Can use online survey technology to complete surveys
* Can download, install and use a smartphone app

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Self-reported 30-day point-prevalence abstinence (PPA) from smoking | Baseline, 2, 6, 12, 24, and 52 weeks
  The 30-day point prevalence abstinence (PPA) is a self-reported measure recorded at 6 months post-quit. In each online survey participant will be asked to report, "During the past 30 days, on how many days did you smoke". If a participant does not report abstinence, they will be asked to indicate how many cigarettes they smoked per day on the days they smoked and whether they are seriously thinking of quitting smoking. The investigators will also include the question, "have you been abstinent during the past 30 days?" (yes/no). In order to get to this question, participants will answer have to answer prior questions as, " I do not smoke at all", and "yes", they have been abstinent during the past 7 days. The investigators will code a binary indicator for self-reported 30-day point prevalence abstinence (yes/ no).

SECONDARY OUTCOMES:
Self-reported 7-day point-prevalence abstinence (PPA) from smoking | Baseline, 2, 6, 12, 24, and 52 weeks
  The investigators will measure 7-day PPA (smoking abstinence) using the same smoking status self-report form described above for 30-day PPA. In each online survey, participants will be asked: "what is your current smoking status?" with the following options: "I smoke daily", "I smoke non-daily (and have smoked in the past 7 days)" , "I smoke non-daily (but have NOT smoked in the past 7 days)" , "I do not smoke at all". If participants have indicated that they do not smoke, they will be asked whether they have been abstinent during the past 7 days (yes/no).
Change in cigarettes smoked | 2, 6, 12, 24, and 52 week after baseline
  In each online survey after the baseline, participants will be asked: "what is your current smoking status?" If a participant does not report abstinence, they will be asked to indicate how many cigarettes they smoked over the past 7 days. The investigators will code an indicator of cigarette reduction by subtracting the total number of cigarettes smoked in the week before baseline from the total number of cigarettes smoked in the past week. Negative change numbers indicate better progress towards smoking cessation.
Smoking self-efficacy | Baseline, 2, 6, 12, 24, and 52 weeks
  A single-item measure that assess a person's confidence in their ability to quit smoking / stay quit will be included. Participants will be asked to rate their answer to the question "How confident are you that you will be able to quit smoking/stay quit?" on a 1-100 slider scale (i.e., 1=not at all confident, 100=absolutely confident). Higher scores indicate greater self-efficacy to abstain from smoking.
Positive affect | Baseline, 2, 6, 12, 24, and 52 weeks
  The investigators will measure positive affect using the Positive and Negative Affect Schedule (PANAS). The PANAS is a 20-item measure assessing intensity with which individuals experience various emotional states in the preceding two weeks, 10 of which assess positive emotional states (e.g., proud) and 10 of which assess negative emotional states (e.g., afraid), on a 1-5 scale (i.e., 1=very slightly or not at all; 5=extremely). Scores for the positive words are summed to yield a positive affect score, with higher scores indicating higher positive affect (positive outcome).
Negative affect | Baseline, week 2, 6, 12, 24, and 52
  The investigators will measure negative affect using the Positive and Negative Affect Schedule (PANAS). The PANAS is a 20-item measure assessing intensity with which individuals experience various emotional states in the preceding two weeks, 10 of which assess positive emotional states (e.g., proud) and 10 of which assess negative emotional states (e.g., afraid), on a 1-5 scale (i.e., 1=very slightly or not at all; 5=extremely). Scores for the negative words are summed to yield a negative affect score, with higher scores indicating higher negative affect (negative outcome).
Mood and Physical Symptoms Scale (MPSS) (modified) | Baseline, 2, 6, 12, 24, and 52 weeks
  The Mood and Physical Symptoms Scale (MPSS) is a cigarette withdrawal scale. The measure focuses on mood and other symptoms of cigarette withdrawal. Items 1-7 list symptoms of withdrawal. Each item is on a scale from 1 ("not at all") to 5 ("extremely") and asked within the in the past 24 hours. The measure also captures the frequency (Item 8; 0, "Not at all" to 5, "All the time") and strength (Item 9; 0, "No urges" to 5, "Extremely strong") of the urge to smoke. The original scale included 12-items, but the investigators only included the first 9 items as being relevant to nondaily smokers. The investigators will use the total of all items (1-9) as a composite score of withdrawal symptoms and urge, where higher scores indicate greater withdrawal and smoking urge (negative outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Hoeppner, Ph.D., M.S., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will provide de-identified IPD related to the aims, baseline demographics, and outcomes described in this study record to interested individuals one year following achievement of the aims of the project (i.e., publication of the main outcome papers). Data sharing will be contingent on meeting all institutional regulations for data use agreements and on receiving evidence of the recipient's institution's IRB approval for planned analyses of the data. The investigator team will be available to address queries.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The investigators will provide de-identified data from this project to interested individuals one year following achievement of the aims of the project (i.e., publication of the main outcome papers).
Access Criteria: Data sharing will be contingent on meeting all institutional regulations for data use agreements and on receiving evidence of the recipient's institution's IRB approval for planned analyses of the data. Interested parties requesting data will receive the requested data needed to execute their analysis plan in accordance with these approvals. The IPD will be provided in digital format with clear labels for all variables, will be de-identified before it is shared, and will be released directly by the investigators to the recipients with secure data tranfer.
  Regarding supporting information, the final version of the study protocol (including the statistical analysis plan (SAP)) and the final version of the Informed Consent Form (ICF) will be made publicly available in this clinicaltrials.gov record. Additional supporting information, including analytic code, will be made available upon a specific request to the investigative team.

REFERENCES:
- [Background] Hoeppner BB, Kelly JF, Urbanoski KA, Slaymaker V. Comparative utility of a single-item versus multiple-item measure of self-efficacy in predicting relapse among young adults. J Subst Abuse Treat. 2011 Oct;41(3):305-12. doi: 10.1016/j.jsat.2011.04.005. Epub 2011 Jun 22. PMID 21700411
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] West R, Hajek P. Evaluation of the mood and physical symptoms scale (MPSS) to assess cigarette withdrawal. Psychopharmacology (Berl). 2004 Dec;177(1-2):195-9. doi: 10.1007/s00213-004-1923-6. Epub 2004 Jun 4. PMID 15179542